CLINICAL TRIAL: NCT02919800
Title: A Phase 1,Randomized, Single-blind, Placebo-controlled, Single Dose, Dose-escalated Study to Assess the Safety, Pharmacokinetic and Pharmacodynamic Profile of Subcutaneous Administration of a Long-acting Recombinant Factor VIIa in Healthy Adult Males
Brief Title: A Single-dose, Dose-escalation Study of a Long-acting MOD-5014 in Healthy Adult Male
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OPKO Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CP-5-002
Record Dates: First submitted 2016-08-11; First posted 2016-09-29 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Hemophilia A or B With Inhibitors
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MOD-5014 (Experimental): MOD-5014 longevity is the result of fusion of three consecutive C-terminal peptide (CTP) domains to the C-terminus of FVII. CTP technology is based on a natural peptide, the C-terminal peptide of the beta chain of human chorionic gonadotropin (hCG), which provides hCG with the required longevity to maintain pregnancy (initial half-life [t1/2] ~10 h, terminal t1/2 ~37 h). The beta chain of luteinizing hormone (LH), a gonadotropin that triggers ovulation, is almost identical to hCG but does not include the CTP. As a result, LH has a significantly shorter half-life in blood (initial t1/2 ~1 h, terminal t1/2 ~10 h) (Fares et al., 1992).
  Interventions: Biological: MOD-5014
- MOD-5014 Placebo (Placebo Comparator): Placebo solution for SC injection containing the same inactive ingredients used in the active drug product at matching volumes
  Interventions: Other: MOD-5014 Placebo

INTERVENTIONS:
Biological: MOD-5014 — MOD-5014, a long-acting modified recombinant Factor VIIa
  Arms: MOD-5014
Other: MOD-5014 Placebo — Placebo solution for SC injection containing the same inactive ingredients used in the active drug product at matching volumes
  Arms: MOD-5014 Placebo

SUMMARY:
A Phase 1, randomized, single-blind, placebo-controlled, single dose, dose-escalation study to assess the safety, pharmacokinetic and pharmacodynamic profile of subcutaneous administration of a long-acting recombinant factor VIIa (MOD-5014) in healthy adult males.

DETAILED DESCRIPTION:
This will be a single-dose, randomized, single-blind, placebo-controlled, dose-escalating study.

The study will include four escalating dose groups, with eight subjects in each dose group. Subjects will be randomized in 3:1 ratio to receive a single SC injection of MOD-5014 (n=6) or a placebo (n=2), and will be followed up for 30 days. The initial MOD-5014 dose group will receive 100 µg/kg followed by single doses of 200, 400 and 600 µg/kg administered to subsequent subject cohorts.

The decision to proceed to the higher dose level will be made by a Data Safety Monitoring Board (DSMB) after review of relevant safety data (including adverse events, clinical laboratory and vital signs), collected up to and including 7 days after the last subject of the previous dose group has been dosed.

Common Terminology Criteria for Adverse Events (CTCAE) guidelines will be used to determine maximum tolerated dose (MTD) and dose limiting toxicity (DLT). Dose escalation will be permitted if the prior dose is well tolerated, and there are no safety or tolerability concerns raised by the investigator, sponsor, medical monitor or DSMB over 7 days post-dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Men, 18-50 years of age, inclusive, at the screening visit.
2. Subjects must provide written informed consent prior to participating in the study.
3. Considered healthy based on medical history, physical examination and clinical laboratory results.
4. Body Mass Index (BMI) 19.0-30.0 kg/m2 and total body weight >50 Kg.
5. Fertile men must agree to use a barrier contraceptive (condom) for 30 days post-dosing and are restricted from donating sperm for 30 days after dosing. Subjects with a vasectomy performed more than 6 months prior to treatment are also acceptable.
6. Supine blood pressure and heart rate within normal limits (systolic 90-140 mmHg; diastolic 50-90 mmHg, heart rate 45-100 beats per minute). No evidence of orthostatic hypotension.
7. Triglyceride ≤ 200 mg/dl
8. ECG with no clinically significant abnormalities recorded at Screening visit and on dosing day (before drug administration): PR interval within 120 and 210 ms, QRS interval < 120 ms, and QTc interval 450 ms.
9. Negative human immunodeficiency virus (HIV), hepatitis B or hepatitis C serology tests at screening.
10. Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
11. Non-smoking and no use of any tobacco or nicotine product by declaration for a period for at least 6 month prior to screening period.

Exclusion Criteria:

1. Family history of blood clots.
2. Have had, within one month prior to study drug administration, a major surgical procedure (e.g. orthopedic, abdominal) or have an elective surgery planned within the study period.
3. Any history of arterial and/or venous thromboembolic events (such as myocardial infarction, ischemic strokes, transient ischemic attacks, deep venous thrombosis or pulmonary embolism).
4. History or current drug/alcohol abuse (excluding use of medicinal cannabis for pain management). History of regular alcohol consumption exceeding - 14 drinks/week for men (1 drink = 5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) within 6 months of screening. Positive urine drug of abuse (DoA) in screening and on admission. Positive breath alcohol test on admission.
5. Known allergy to any drug. Known allergy or hypersensitivity to any of the test compounds or materials or contraindication to test product.
6. Use of any prescription or over-the-counter (OTC) medications, including vitamins and herbal or dietary supplements within 14 days prior to dosing. Paracetamol for symptomatic relief of pain is allowed until 24 hours prior to the study drug administration.
7. Subjects who have received any vaccines within 4 weeks prior to study drug administration.
8. Participation in another clinical trial within 30 days.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2017-01-22 (Actual); Primary Completion 2018-02-21 (Actual); Study Completion 2018-02-21 (Actual)

PRIMARY OUTCOMES:
Composite safety and tolerability parameters as measured by adverse events, electrocardiograms (ECG), Immunogenicity, laboratory results, vital signs and injection site reactions | within 30 days of injection

SECONDARY OUTCOMES:
Cmax of MOD-5014 | within 30 days of injection
Tmax of MOD-5014 | within 30 days of injection
AUC(0-t) of MOD-5014 | within 30 days of injection
AUC(inf) of MOD-5014 | within 30 days of injection
T(½) of MOD-5014 | within 30 days of injection
Clearance of MOD-5014 | within 30 days of injection

CONTACTS AND LOCATIONS:
Overall Officials: Ramit Arison, Study Director — Associate Director Clinical Affairs OPKO Biologics
Locations (1):
- TASMC, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bysted BV, Scharling B, Moller T, Hansen BL. A randomized, double-blind trial demonstrating bioequivalence of the current recombinant activated factor VII formulation and a new robust 25 degrees C stable formulation. Haemophilia. 2007 Sep;13(5):527-32. doi: 10.1111/j.1365-2516.2007.01516.x. PMID 17880439
- [Result] Fares FA, Suganuma N, Nishimori K, LaPolt PS, Hsueh AJ, Boime I. Design of a long-acting follitropin agonist by fusing the C-terminal sequence of the chorionic gonadotropin beta subunit to the follitropin beta subunit. Proc Natl Acad Sci U S A. 1992 May 15;89(10):4304-8. doi: 10.1073/pnas.89.10.4304. PMID 1374895
- [Result] Fridberg MJ, Hedner U, Roberts HR, Erhardtsen E. A study of the pharmacokinetics and safety of recombinant activated factor VII in healthy Caucasian and Japanese subjects. Blood Coagul Fibrinolysis. 2005 Jun;16(4):259-66. doi: 10.1097/01.mbc.0000169218.15926.34. PMID 15870545
- [Result] Klitgaard T, Nielsen TG. Overview of the human pharmacokinetics of recombinant activated factor VII. Br J Clin Pharmacol. 2008 Jan;65(1):3-11. doi: 10.1111/j.1365-2125.2007.03030.x. Epub 2007 Oct 24. PMID 17961193
- [Result] Moss J, Scharling B, Ezban M, Moller Sorensen T. Evaluation of the safety and pharmacokinetics of a fast-acting recombinant FVIIa analogue, NN1731, in healthy male subjects. J Thromb Haemost. 2009 Feb;7(2):299-305. doi: 10.1111/j.1538-7836.2008.03253.x. Epub 2008 Dec 3. PMID 19138379
- [Result] Tanaka KA, Key NS, Levy JH. Blood coagulation: hemostasis and thrombin regulation. Anesth Analg. 2009 May;108(5):1433-46. doi: 10.1213/ane.0b013e31819bcc9c. PMID 19372317